CLINICAL TRIAL: NCT04192071
Title: Adapting and Pilot Testing a Nutrition Module Delivered With Virtual Human Technology for Colorectal Cancer Prevention
Brief Title: Virtual Human Delivered Nutrition Module for Colorectal Cancer Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: IRB201902537; 3R01CA207689-03S2 (NIH); OCR27722 (Other: UF OnCore); IRB201902537 (Other: IRB)
Record Dates: First submitted 2019-12-06; First posted 2019-12-10 (Actual); Results first posted 2024-08-28 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Colorectal Cancer
Keywords: Nutrition
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- high interactive virtual human administered nutrition module (Active Comparator): The virtual health assistant will interactively collect nutrition information (alcohol, red meat, and processed meat intake) and report risk information back to users in visual and audio format
  Interventions: Other: virtual technology - high interactive
- low interactive virtual human module (Active Comparator): Complete the current intervention module that includes items assessing alcohol and meat intake.
  Interventions: Other: virtual technology - low interactive
- attention control module (Sham Comparator): The attention control group, will complete a related module not related to colorectal cancer or nutrition
  Interventions: Other: non-colorectal cancer related module

INTERVENTIONS:
Other: virtual technology - high interactive — Participants engage with web-based cancer prevention content and answer a short series of questions designed to assess their baseline risk for colon cancer and dietary intake. Interactive nutrition risk feedback will be customized based on user input.
  Other Names: Virtual human nutrition module
  Arms: high interactive virtual human administered nutrition module
Other: virtual technology - low interactive — Participants engage with web-based cancer prevention content and answer a short series of questions designed to assess their baseline risk for colon cancer. Minimally interactive risk feedback will be delivered.
  Other Names: virtual human standard
  Arms: low interactive virtual human module
Other: non-colorectal cancer related module — Participants engage with web-based content not related to colorectal cancer or nutrition.
  Other Names: attention control
  Arms: attention control module

SUMMARY:
This study uses the opinions of adults between the ages of 45 and 73 years old to develop and test an interactive nutrition module for use in an existing colorectal cancer screening intervention using virtual human technology. The main questions answered include:

* What content do adults want to receive from a web-based interaction about colorectal cancer screening and nutritional risks for colorectal cancer?
* Does a brief interaction with a virtual human delivering tailored cancer prevention information impact cancer prevention intentions and attitudes among a national sample of geographically rural U.S. adults?

This study will contribute to knowledge of what messages and graphics promote understanding of cancer risk and promote screening with the potential to promote behaviors that reduce cancer risk.

DETAILED DESCRIPTION:
The study occurred in two phases. Phase one was a qualitative aim that collected feedback from participants in iterative cycles of focus groups and individual think-aloud interviews. Phase one feedback was analyzed and applied to develop a tailored, web-based prototype that addressed participant desires for an intervention to address colorectal cancer prevention and nutrition risk education. The prototype was a brief conversation delivered by an interactive Virtual Health Assistant (virtual character with audio and visual elements that mimic a conversation with a human).

ELIGIBILITY:
Inclusion Criteria:

* Eligible adults will be between 45 -73 years old,
* Proficient in English and
* Geographically residing in rural areas (based on zip code)
* Identify as Black or White racial identity

Exclusion:

* Completed a colonoscopy in the past 10 years
* Completed a sigmoidoscopy in the past 5 years
* Completed a home stool test in the past 12 months

Ages: 45 Years to 73 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2022-06-27 (Actual); Study Completion 2022-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Vilaro, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vilaro MJ, Bryan E, Palani T, Cooks EJ, Mertens G, Zalake M, Lok BC, Krieger JL. Rural adults' perceptions of nutrition recommendations for cancer prevention: Contradictory and conflicting messages. Prev Oncol Epidemiol. 2023;1(1):2237680. doi: 10.1080/28322134.2023.2237680. Epub 2023 Nov 17. PMID 38390218
- [Result] Vilaro MJ, McAlindon K, Mertens G, Ashley T, Zalake M, Cooks EJ, Krieger JL. Information Architects: Using Community-Engaged and Qualitative Methods to Design a Technology-Based Nutrition and Cancer Risk Intervention for Rural Adults. Cancer Control. 2023 Jan-Dec;30:10732748221130162. doi: 10.1177/10732748221130162. PMID 36919704

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Aim 2 Pilot Test: Web-based, single-interaction, intervention Aim 2 intervention development (focus groups and interviews)
Pre-assignment Details: Total N =139 (Aim 1 = 48; Aim 2 = 91)
  AIMS 1 & 2 are independent. Aim 1 participants did NOT complete Aim 2.
  (AIM 2) Qualtrics panels recruited a national sample of (n=91) rural adults. Respondents from this national sample who did not meet the qualifying criteria were screened out by the Qualtrics platform and did not get randomized to one of the 3 arms of the web-based, intervention.
  ( AIM 1) participants (n=48) completed focus groups/interviews informing intervention content.
Groups:
- AIM 1 Focus Group and Interview Participants: a total of 48 participants completed focus groups and interviews to provide feedback on iteratively updated versions of the culturally tailored, web-based, intervention, and participate in user testing. These participants did NOT participate in the AIM 2 pilot testing of the 3-arm, randomized trial.
Period: Overall Study
Arm/Group | High Interactive Virtual Human Administered Nutrition Module | Low Interactive Virtual Human Module | Attention Control Module | AIM 1 Focus Group and Interview Participants
Started | 31 | 35 | 25 | 48
Completed | 31 | 35 | 25 | 48
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Aim 2 Web-based Pilot Test: Control: participants interact with attention control information about clinical trials (not focused on cancer, not focused on nutrition)
- Aim 2 Web-based Pilot Test: Low Interactive Condition: Participants interact with nutrition and cancer risk information in a low interactive condition.
- Aim 2 Web-based Pilot Test: VHA High Interactive Condition: Participants interact with nutrition and cancer risk information delivered by a Virtual Health Assistant in a high interactive condition.
- Aim 1: Focus Group and Interviews: Participants provided feedback to inform the web-based intervention that would be pilot-tested in Aim 2.
- Total: Total of all reporting groups
Arm/Group | Aim 2 Web-based Pilot Test: Control | Aim 2 Web-based Pilot Test: Low Interactive Condition | Aim 2 Web-based Pilot Test: VHA High Interactive Condition | Aim 1: Focus Group and Interviews | Total
Number analyzed (Participants) | 25 | 35 | 31 | 48 | 139
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 21 | 32 | 23 | 31 | 107
  >=65 years | 4 | 3 | 8 | 17 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (8) | 55.1 (7.7) | 57 (9.2) | 61.7 (7) | 56 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 24 | 21 | 24 | 85
  Male | 9 | 11 | 10 | 24 | 54
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 2 | 0 | 3
  Not Hispanic or Latino | 25 | 34 | 29 | 48 | 136
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 12 | 15 | 13 | 31 | 71
  White | 13 | 20 | 18 | 17 | 68
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 25 | 35 | 31 | 48 | 91

OUTCOME MEASURES:

1. Primary Outcome: Risk Perceptions for Colorectal Cancer
Description: Items measured on a 7-point Likert scale, (e.g. "My chances of getting colorectal cancer are high"), where 1 is strongly disagree and 7 is strongly agree.
Time Frame: up to 2 hours
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Aim 2 Web-based Pilot Test: Control | Aim 2 Web-based Pilot Test: Low Interactive Condition | Aim 2 Web-based Pilot Test: VHA High Interactive Condition
Number analyzed (Participants) | 25 | 35 | 31
score on a scale | 3.3 (1.5) | 3.6 (1.4) | 3.5 (1.3)

2. Primary Outcome: Intentions to Screen for Colorectal Cancer
Description: Two individual items assessed intentions to screen:
  1. A single item measured intentions to screen for colorectal cancer (readiness to screen) adapted from (Boonyasiriwat, Hung, Hon, et. al, 2014.) Participants answer the following prompt: "Please indicate what best represents your plans for colorectal cancer screening". Response options str: 1 point = I am not planning to screen in the next 6 months; 2 points = I am thinking about screen, but not in the next 6 months; 3 points = I am considering screening in the next 6 months and 4 points for = I am already taking steps to screen in the next 6 months. Higher scores =higher readiness to screen (better outcome). Min. score = 1 ; Max. score =4.
  2. a single item assessed intentions on a Likert Scale. Question: "I want to get screened for colorectal cancer" where: 1 = strongly disagree-7 = strongly agree). Min. score = 1 - Max. score is 7. Higher scores indicate a stronger desire to obtain screening (better outcome).
Time Frame: up to 2 hours
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Aim 2 Web-based Pilot Test: Control | Aim 2 Web-based Pilot Test: Low Interactive Condition | Aim 2 Web-based Pilot Test: VHA High Interactive Condition
Number analyzed (Participants) | 25 | 35 | 31
score on a scale
  4 point, 6-month readiness | 2.6 (1) | 2.5 (1) | 2.5 (.8)
  7-point Likert Intention | 5 (1.6) | 4.9 (2.0) | 5.2 (1.4)

3. Primary Outcome: Information Seeking Behavior
Description: Does participant click on link to more information. The survey platforms event tracking feature will be used to track clicks (yes/no) for more information.
Time Frame: up to 2 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Aim 2 Web-based Pilot Test: Control | Aim 2 Web-based Pilot Test: Low Interactive Condition | Aim 2 Web-based Pilot Test: VHA High Interactive Condition
Number analyzed (Participants) | 25 | 35 | 31
Participants
  No | 11 | 14 | 14
  Yes | 14 | 21 | 17

ADVERSE EVENTS:
Time Frame: We did not monitor adverse events as the potential risks were not more than would be expected in every day life. There are no potential risks of physical, psychological or economic harm associated with participating in this study.
Description: Participants engaged in focus groups, interviews and remote completion of a one-time, web-based educational interaction, thus we did not collect adverse events.
Groups:
- Aim 1 Focus Groups and Interviews: Participants provided feedback to inform the iterative development of web-based colorectal cancer and nutrition risk interaction with a virtual health assistant.
Arm/Group | Aim 2 Web-based Pilot Test: Control | Aim 2 Web-based Pilot Test: Low Interactive Condition | Aim 2 Web-based Pilot Test: VHA High Interactive Condition | Aim 1 Focus Groups and Interviews
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2022-05-24): https://cdn.clinicaltrials.gov/large-docs/71/NCT04192071/Prot_SAP_000.pdf
  • Informed Consent Form: Pilot test (2022-02-15): https://cdn.clinicaltrials.gov/large-docs/71/NCT04192071/ICF_001.pdf
  • Informed Consent Form: Think aloud (2020-10-05): https://cdn.clinicaltrials.gov/large-docs/71/NCT04192071/ICF_002.pdf